CLINICAL TRIAL: NCT00166023
Title: A Review of Outcomes Following Medical or Surgical Management of Endocarditis
Brief Title: Outcomes Following Medical or Surgical Management of Endocarditis
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Brian Kogon, Principal Investigator, Emory University
Other Study IDs: 0549-2005
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2013-11-26 (Estimated); Status verified 2013-11

CONDITIONS: Endocarditis
Keywords: pediatric; cardiology
MeSH Terms: conditions — Endocarditis

SUMMARY:
Infective endocarditis is a rare disease, and while there have been several large reviews of the incidence of endocarditis in the pediatric patient population, relatively little has been published regarding the short and medium-term outcomes following medical and surgical therapy for this disease. The goal is to compare the outcome for children treated for endocarditis with either medical management or surgery by looking at the success of these two treatment strategies. Another goal is to attempt to identify risk factors for medical management that might identify patients who would be better served by early surgery.

DETAILED DESCRIPTION:
After identification of qualified subjects, the families of surviving patients will be mailed a package containing a cover letter explaining the study, a consent form, an assent form if applicable, a questionnaire (designed to evaluate longer-term outcome measures including the occurrence of recurrent endocarditis, late surgical intervention or the need for re-operations) and a self addressed stamped envelope to be used to return the consents and the questionnaire. The data will then be entered into a database and analyzed.

ELIGIBILITY:
Inclusion Criteria:

* All patients discharged from Children's Healthcare of Atlanta at Egleston with a discharge diagnosis of endocarditis or those who underwent surgery with a preoperative diagnosis of endocarditis.
* Admitted to the hospital between January 1, 1984 - December 31, 2004, inclusive.
* Signed informed consent.

Exclusion Criteria:

* Patients who do not have documented endocarditis based upon microbiology and echocardiography criteria.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 2005-08; Study Completion 2006-12

CONTACTS AND LOCATIONS:
Overall Officials: Paul Kirshbom, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States